CLINICAL TRIAL: NCT06988059
Title: A Clinical Study to Explore the Safety, Efficacy, and Pharmacokinetics of CT0596 CAR-T Cell Injection in Patients With Plasma Cell Leukemia
Brief Title: A Study of CT0596 in Plasma Cell Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025050
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Plasma Cell Leukemia
Keywords: Plasma Cell Leukemia; CAR-T cells
MeSH Terms: conditions — Leukemia, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T cells Infusion chimeric antigen receptor T cells (Experimental)
  Interventions: Drug: CAR-T cells Infusion chimeric antigen receptor T cells

INTERVENTIONS:
Drug: CAR-T cells Infusion chimeric antigen receptor T cells — CAR-T cells Infusion

SUMMARY:
This study is a single-arm, open-label, exploratory dose-escalation and dosefinding clinical trial to evaluate the safety, efficacy, cellular pharmacokinetics and pharmacodynamics of CT0596 cells in patients with PCL.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, exploratory dose-escalation and dosefinding clinical trial to evaluate the safety, efficacy, cellular pharmacokinetics and pharmacodynamics of CT0596 cells in patients with PCL. During the trial, dose increases or decreases or dose expansion may be performed using i3+3 principle based on the safety and ,tolerability and PK data of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must voluntarily sign the informed consent form (ICF) and must be willing and be able to adhere to the trial visit schedule and other protocol requirements and agree to be in long term follow-up (LTFU) for up to 15 years as mandated by the regulatory guidelines.
2. Age ≥ 18 years;
3. PCL after inductive treatment or R/R pPCL.
4. Patients must have measurable disease。
5. Expected survival > 12 weeks;
6. Eastern Cooperative Oncology Group (ECOG) score 0- 1 ;
7. Patients should have good organ function。
8. Female patients of childbearing potential must have a negative pregnancy test at screening and prior to receiving lymphodepletion therapy and are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment and are absolutely prohibited from donating eggs for 1 year after receiving study treatment infusion during the study ;Male patients are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment if they are sexually active with a female of childbearing potential. Sperm donation is absolutely prohibited within 1 year following study treatment infusion for all male patients during the study.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients seropositive for HIV, active hepatitis C virus (HCV), or active hepatitis B virus (HBV) infection. History of treated hepatitis B or C is permitted if the viral load is undetectable per qPCR and or nucleic acid testing;
3. Patients with any uncontrolled active infection, including but not limited to patients with active tuberculosis (investigator 's judgment);
4. Toxicities caused by previous treatment have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade 1, except alopecia and other events that are judged tolerable by the investigator;
5. Patient has any significant condition(s), laboratory abnormality or psychiatric illness that would impair the ability of the patient to receive or tolerate the planned treatment or in the opinion of the investigator, participation would not be in the best interest of the patient (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
6. Previous allogeneic stem cell transplantation; autologous stem cell transplantation within 12 weeks prior to signing informed consent;
7. Have received treatment for the disease within 14 days or five half-lives before preconditioning
8. Have received cell therapy within 28 days before informed consent.
9. Systemic glucocorticoids equivalent to > 15 mg/day prednisone within 7 days prior to informed consent, with the exception of topical glucocorticoids;
10. Vaccination with live attenuated vaccines , inactivated vaccines or RNA vaccines within 4 weeks prior to informed consent;
11. Major surgery within 2 weeks before informed consent or planned during the study period or within 4 weeks after giving study treatment (excluding local anesthesia such as cataract);
12. Allergic or intolerant to lymphodepletion, tocilizumab, or allergic to components (DMSO) in CT0596 CART cell infusion preparation; or previous history of other serious allergies such as anaphylactic shock;
13. Patients with secondary plasma cell leukemia, Waldenström macroglobulinemia, POEMS syndrome, or primary light chain amyloidosis at screening;
14. Patients with any of the following cardiac conditions within 6 months prior to screening:
15. Patients who require supplemental oxygen to maintain oxygen saturation > 92%; or Patients with known or suspected COPD who have Forced Expiratory Volume in 1 second (FEV1) < 50% of predicted normal on spirometry;
16. Patients with active autoimmune diseases, including but not limited to psoriasis, rheumatoid arthritis and other diseases requiring long-term immunosuppressive therapy;
17. Patients with second primary malignancies in addition to MM are not eligible if the second primary malignancy has required treatment within the past 2 years or is not in complete remission. Exceptions include the following that have been successfully treated - nonmetastatic basal cell or squamous cell skin carcinoma, non-metastatic prostate cancer, carcinoma-in-situ of breast or cervix, non-muscle invasive bladder cancer
18. Patients with symptomatic central nervous system (CNS) disease or suspected CNS metastases;
19. The patient is unable or unwilling to comply with protocol, or there are other reasons for being unsuitable to participate in this clinical study evaluated by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-01-03 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) after CT0596 infusion | 12 months after CT0596 infusion
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria
MTD and/or dose range | 12 months after CT0596 infusion
  Evaluate Dose limited toxicity and recommended dosage range after CT0596 infusion

SECONDARY OUTCOMES:
Overall response rate (ORR) as assessed by the investigator | 12 months after CT0596 infusion
  Overall response rate (ORR) defined as proportion of patients achieving partial response or better based on International Myeloma Working Group defined response criteria
Complete response/stringent complete response (CR/sCR) rate | 12 months after CT0596 infusion
  Rate of complete response/stringent complete response (CR/sCR) defined as proportion of patients achieving CR or better based on IMWG defined response criteria.
Rate of very good partial response (VGPR) and above | 12 months after CT0596 infusion
  Rate of complete very good partial response response/stringent complete response (VGPR/CR/sCR) defined as proportion of patients achieving VGPR or better based on IMWG defined response criteria
Duration of response (DOR) | 12 months after CT0596 infusion
  DOR is defined as the time from first achieving PR or better to confirmed disease progression or death from any cause
Minimal residual disease (MRD) negative rate | 12 months after CT0596 infusion
  Minimal residual disease (MRD) negative rate is defined as the proportion of patients with VGPR or better who achieved 10-5 sensitivity of nucleated cell
Time to response (TTR) | 12 months after CT0596 infusion
  TTR defined as the time from the date of infusion to the date of initial assessment of PR or better according to IMWG2016 criteria
Progression-free survival (PFS) | 12 months after CT0596 infusion
  PFS defined as the time from the date of infusion of the subject to the first assessment of confirmed disease progression or death from any cause according to IMWG2016 criteria, whichever occurs first.
Peak value of CART cells | 12 months after CT0596 infusion
  Time to peak expansion and peak expansion in plasma after infusion of CT0596 cells
Overall survival (OS) | 12 months after CT0596 infusion
  OS defined as the time from the date of infusion of the subject to death from any cause
Cytokines in the peripheral blood after CT0596 infusion | 12 months after CT0596 infusion
  Serum concentrations of interleukin (IL)-6 after CT0596 infusion
Area under the plasma concentration versus time curve (AUC) of CART cells | 12 months after CT0596 infusion
  Area under the plasma concentration versus time curve (AUC) in plasma after infusion of CT0596 cells
In vivo persistence of CART cells | 12 months after CT0596 infusion]
  CART cells duration in plasma after infusion of CT0596 cells

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No